CLINICAL TRIAL: NCT01660126
Title: Multi-modal Effects of Thyroid Hormone Replacement for Untreated Older Adults With Subclinical Hypothyroidism; a Randomised Placebo-controlled Trial
Brief Title: Thyroid Hormone Replacement for Subclinical Hypothyroidism
Acronym: TRUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); University College Cork (Other); University of Bern (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Professor David J Stott, David Cargill Professor of Geriatric Medicine, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN11GE272; 2011-004554-26 (EudraCT Number)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Subclinical Hypothyroidism
Keywords: Aged; Cardiovascular disease; Levothyroxine; Randomised controlled trial; Quality of life; Subclinical hypothyroidism
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levothyroxine (Active Comparator): Oral Levothyroxine, starting dose 25 or 50 micrograms increased to a maximum of 150 micrograms once daily.
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — The intervention will start with Levothyroxine 50 µg daily (reduced to 25 µg in subjects <50Kg body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) versus matching placebo; at 3 months if the serum TSH level is <0.4 mU/L dose will be reduced by 25 µg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6mUL, additional 25 µg. The process will be repeated at 12 months then annually. Mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine that will be prescribed is 150μg.
  Other Names: Thyroxine
  Arms: Levothyroxine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Subclinical hypothyroidism (SCH) is a common condition among older men and women. Although by definition SCH comprises biochemically mild thyroid hormone deficiency without overt symptoms, it is a possible contributor to multiple problems in older age. Thyroid hormone has effects on numerous physiological systems, including the vascular tree, heart, skeletal muscle and brain. Therefore, thyroxine substitution to overcome thyroid hormone deficiency has the potential to give multisystem benefits to older people with SCH.

Small studies have reported reduced atherosclerosis and improved heart function with thyroxine replacement, but no large clinical trials have been performed. Therefore the available evidence is limited, leading to major variations in guidelines and clinical practice, with uncertainty regarding the indications for screening and treatment. The investigators propose a multicentre randomised placebo controlled trial to assess the impact of thyroxine replacement in a minimum of 540 older adults (maximum 750) with persisting SCH (excluding those in whom it is a temporary phenomenon who are unlikely to benefit). The investigators will include older men and women with a wide age range and of varying health status. Outcomes include health related quality of life, muscle strength, executive cognitive function and cardiovascular events, with a minimum of 1 year of follow up. Blood and urine samples will be stored in a biobank, to allow future research on causes of ill health in older people with SCH.

The investigators have the support of patient advocacy groups and a consortium with the wide range of expertise and experience required to conduct large scale multicentre clinical trials. The proposal explores the multisystem and quality of life benefits to older people of a tailored approach to management of SCH.

This clinical trial should definitively clarify whether thyroxine treatment for SCH provides benefits that are relevant for patients. This trial will provide strong evidence with the potential to improve clinical practice, reduce health care costs and promote healthy ageing of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients aged >=65 years with Subclinical Hypothyroidism (SCH).

SCH is defined as elevated TSH levels (>=4.6, <=19.9 mU/L) and free thyroxine (fT4) in reference range measured on a minimum of two occasions at least 3 months apart.

Exclusion Criteria:

* Subjects currently on Levothyroxine or antithyroid drugs, amiodarone or lithium.
* Recent thyroid surgery or radio-iodine (within 12 months).
* Grade IV NYHA heart failure.
* Prior clinical diagnosis of dementia.
* Recent hospitalisation for major illness or elective surgery (within 4 weeks).
* Recent acute coronary syndrome, including myocardial infarction or unstable angina (within 4 weeks).
* Terminal illness.
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Subjects who are participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Plan to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 737 (Actual)
Dates: Start 2014-05; Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Thyroid-specific quality of life - Hypothyroid symptoms and Fatigue symptoms (co-primary outcomes) | Measured at baseline and 12 months
  Change in Hypothyroid Symptoms and Fatigue scores (measured using the Thyroid-specific quality of life Patient Reported Outcome questionnaire - ThyPRO; Hypothyroid symptoms and Fatigue domains).

SECONDARY OUTCOMES:
Health-related quality of life | measured at baseline; 3 month; 12 month and final follow up (expected mean follow-up of 18 months).
  The EuroQol5D
Handgrip strength | Measured at baseline; 12 months and final follow up (expected mean follow-up of 18 months).
  Handgrip strength measured using the Jadaar hand dynamometer.
Executive cognitive function | Measured at baseline and final follow-up (expected mean follow-up of 18 months).
  Letter Digit Coding Test [LDCT).
Total mortality | Up to final follow up (expected mean follow-up of 18 months).
  Total mortality
Basic Activities of Daily Living | Measured at baseline and final follow-up (expected mean follow-up of 18 months).
  Basic Activities of Daily Living (ADL) measured using the 20-point Barthel Index [BI].
Extended activities of daily living | Measured at baseline and final follow-up (expected mean follow-up of 18 months).
  Extended activities of daily living measured using the older American resources and services [OARS]) questionnaire
Haemoglobin | Measured at baseline and 1 year
  Change in haemoglobin, measured on a full blood count
Fatal and non-fatal cardiovascular events | Expected mean follow-up of 18 months.
  This will include fatal and non fatal acute myocardial infarction and stroke; amputations for peripheral vascular disease; revascularisations for atherosclerotic vascular disease, including for acute coronary syndrome; heart failure hospitalisations.
Generic thyroid specific quality of life | Final follow-up
  Thyroid-related quality of life Patient-Reported Outcome measure (ThyPRO) 39
Thyroid-specific quality of life - Hypothyroid symptoms | Measured at 6-8 weeks and at final review
  Change in hypothyroid symptom burden (measured using the Thyroid-specific quality of life Patient Reported Outcome questionnaire - ThyPRO; Hypothyroid symptoms domain).
Thyroid specific quality of life - Fatigue symptoms | Measured at 6-8 weeks and at final review
  Change in fatigue (measured using the Thyroid-specific quality of life Patient Reported Outcome questionnaire - ThyPRO; Fatigue and vitality domain).

CONTACTS AND LOCATIONS:
Overall Officials: David J Stott, MBChB MD, Principal Investigator — University of Glasgow; Jacobijn Gussekloo, MD, Principal Investigator — Leiden University Medical Center; Nicolas Rodondi, MD, Principal Investigator — University of Bern; Patricia Kearney, MD, Principal Investigator — University College Cork; Rudi JG Westendorp, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Glasgow Royal Infirmary, NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

REFERENCES:
- [Derived] van der Spoel E, van Vliet NA, Poortvliet RKE, Du Puy RS, den Elzen WPJ, Quinn TJ, Stott DJ, Sattar N, Kearney PM, Blum MR, Alwan H, Rodondi N, Collet TH, Westendorp RGJ, Ballieux BE, Jukema JW, Dekkers OM, Gussekloo J, Mooijaart SP, van Heemst D. Incidence and Determinants of Spontaneous Normalization of Subclinical Hypothyroidism in Older Adults. J Clin Endocrinol Metab. 2024 Feb 20;109(3):e1167-e1174. doi: 10.1210/clinem/dgad623. PMID 37862463
- [Derived] Netzer S, Chocano-Bedoya P, Feller M, Janett-Pellegri C, Wildisen L, Buchi AE, Moutzouri E, Gonzalez Rodriguez E, Collet TH, Poortvliet RKE, Mc Carthy VJC, Aeberli D, Aujesky D, Westendorp R, Quinn TJ, Gussekloo J, Kearney PM, Mooijaart S, Bauer DC, Rodondi N. The effect of thyroid hormone therapy on muscle function, strength and mass in older adults with subclinical hypothyroidism-an ancillary study within two randomized placebo controlled trials. Age Ageing. 2023 Jan 8;52(1):afac326. doi: 10.1093/ageing/afac326. PMID 36721961
- [Derived] Buchi AE, Feller M, Netzer S, Blum MR, Gonzalez Rodriguez E, Collet TH, Del Giovane C, van Heemst D, Quinn T, Kearney PM, Westendorp RGJ, Gussekloo J, Mooijaart SP, Hans D, Bauer DC, Rodondi N, Aeberli D. Bone geometry in older adults with subclinical hypothyroidism upon levothyroxine therapy: A nested study within a randomized placebo controlled trial. Bone. 2022 Aug;161:116404. doi: 10.1016/j.bone.2022.116404. Epub 2022 Apr 2. PMID 35381390
- [Derived] Du Puy RS, Poortvliet RKE, Mooijaart SP, Stott DJ, Quinn T, Sattar N, Westendorp RGJ, Kearney PM, McCarthy VJC, Byrne S, Rodondi N, Baretella O, Collet TH, van Heemst D, Dekkers OM, Jukema JW, Smit JWA, Gussekloo J, den Elzen WPJ. No Effect of Levothyroxine on Hemoglobin in Older Adults With Subclinical Hypothyroidism: Pooled Results From 2 Randomized Controlled Trials. J Clin Endocrinol Metab. 2022 May 17;107(6):e2339-e2347. doi: 10.1210/clinem/dgac106. PMID 35218666
- [Derived] Zijlstra LE, Jukema JW, Westendorp RGJ, Du Puy RS, Poortvliet RKE, Kearney PM, O'Keeffe L, Dekkers OM, Blum MR, Rodondi N, Collet TH, Quinn TJ, Sattar N, Stott DJ, Trompet S, den Elzen WPJ, Gussekloo J, Mooijaart SP. Levothyroxine Treatment and Cardiovascular Outcomes in Older People With Subclinical Hypothyroidism: Pooled Individual Results of Two Randomised Controlled Trials. Front Endocrinol (Lausanne). 2021 May 20;12:674841. doi: 10.3389/fendo.2021.674841. eCollection 2021. PMID 34093444
- [Derived] de Montmollin M, Feller M, Beglinger S, McConnachie A, Aujesky D, Collet TH, Ford I, Gussekloo J, Kearney PM, McCarthy VJC, Mooijaart S, Poortvliet RKE, Quinn T, Stott DJ, Watt T, Westendorp R, Rodondi N, Bauer DC. L-Thyroxine Therapy for Older Adults With Subclinical Hypothyroidism and Hypothyroid Symptoms: Secondary Analysis of a Randomized Trial. Ann Intern Med. 2020 Jun 2;172(11):709-716. doi: 10.7326/M19-3193. Epub 2020 May 5. PMID 32365355
- [Derived] Gonzalez Rodriguez E, Stuber M, Del Giovane C, Feller M, Collet TH, Lowe AL, Blum MR, van Vliet NA, van Heemst D, Kearney PM, Gussekloo J, Mooijaart S, Westendorp RGJ, Stott DJ, Aeberli D, Bauer DC, Hans D, Rodondi N. Skeletal Effects of Levothyroxine for Subclinical Hypothyroidism in Older Adults: A TRUST Randomized Trial Nested Study. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz058. doi: 10.1210/clinem/dgz058. PMID 31702015
- [Derived] Mooijaart SP, Du Puy RS, Stott DJ, Kearney PM, Rodondi N, Westendorp RGJ, den Elzen WPJ, Postmus I, Poortvliet RKE, van Heemst D, van Munster BC, Peeters RP, Ford I, Kean S, Messow CM, Blum MR, Collet TH, Watt T, Dekkers OM, Jukema JW, Smit JWA, Langhorne P, Gussekloo J. Association Between Levothyroxine Treatment and Thyroid-Related Symptoms Among Adults Aged 80 Years and Older With Subclinical Hypothyroidism. JAMA. 2019 Nov 26;322(20):1977-1986. doi: 10.1001/jama.2019.17274. PMID 31664429
- [Derived] Stott DJ, Rodondi N, Kearney PM, Ford I, Westendorp RGJ, Mooijaart SP, Sattar N, Aubert CE, Aujesky D, Bauer DC, Baumgartner C, Blum MR, Browne JP, Byrne S, Collet TH, Dekkers OM, den Elzen WPJ, Du Puy RS, Ellis G, Feller M, Floriani C, Hendry K, Hurley C, Jukema JW, Kean S, Kelly M, Krebs D, Langhorne P, McCarthy G, McCarthy V, McConnachie A, McDade M, Messow M, O'Flynn A, O'Riordan D, Poortvliet RKE, Quinn TJ, Russell A, Sinnott C, Smit JWA, Van Dorland HA, Walsh KA, Walsh EK, Watt T, Wilson R, Gussekloo J; TRUST Study Group. Thyroid Hormone Therapy for Older Adults with Subclinical Hypothyroidism. N Engl J Med. 2017 Jun 29;376(26):2534-2544. doi: 10.1056/NEJMoa1603825. Epub 2017 Apr 3. PMID 28402245
- [Derived] Stott DJ, Gussekloo J, Kearney PM, Rodondi N, Westendorp RG, Mooijaart S, Kean S, Quinn TJ, Sattar N, Hendry K, Du Puy R, Den Elzen WP, Poortvliet RK, Smit JW, Jukema JW, Dekkers OM, Blum M, Collet TH, McCarthy V, Hurley C, Byrne S, Browne J, Watt T, Bauer D, Ford I. Study protocol; Thyroid hormone Replacement for Untreated older adults with Subclinical hypothyroidism - a randomised placebo controlled Trial (TRUST). BMC Endocr Disord. 2017 Feb 3;17(1):6. doi: 10.1186/s12902-017-0156-8. PMID 28158982